CLINICAL TRIAL: NCT03736603
Title: The PIPA Study (Pathways for Improving Pediatric Asthma Care): A Cluster Randomized Trial
Brief Title: Implementing Pathways to Improve Pediatric Asthma Care
Acronym: PIPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Academy of Pediatrics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17 KA 01
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pathway Intervention 1 (Experimental): Hospitals randomized to group 1 receive PIPA Intervention Bundle 1.
  Interventions: Behavioral: PIPA Intervention Bundle 1
- Pathway Intervention 2 (Experimental): Hospitals randomized to group 2 receive PIPA Intervention Bundle 2, which adds a mobile app.
  Interventions: Behavioral: PIPA Intervention Bundle 2
- Control (No Intervention): Hospitals are in the control arm (usual care) after January 2017 until active implementation begins, which includes 3-6 months of implementation preparation (identifying local multidisciplinary champions, educational sessions/webinars for local champions, one teleconference with an external practice facilitator).

INTERVENTIONS:
Behavioral: PIPA Intervention Bundle 1 — The PIPA intervention bundle 1 includes:
  1. Pathway Implementation Toolkit
  2. Local Multidisciplinary Champions
  3. Audit and Feedback
  4. Educational Seminars/Webinars
  5. Practice Facilitation
  Arms: Pathway Intervention 1
Behavioral: PIPA Intervention Bundle 2 — The PIPA intervention bundle 2 includes:
  1. Pathway Implementation Toolkit
  2. Local Multidisciplinary Champions
  3. Audit and Feedback
  4. Educational Seminars/Webinars
  5. Practice Facilitation
  6. Mobile App
  Arms: Pathway Intervention 2

SUMMARY:
Background:

Asthma affects nearly 10% of American children, and is a leading cause of pediatric emergency visits and hospitalizations. Clinical pathways are operational versions of practice guidelines aimed at the hospital management of common illnesses. Single-site studies of pediatric asthma pathways have shown significant improvements in quality of care.

Primary Objective:

To evaluate the effectiveness of clinical pathways for improving quality of care for children with asthma in a diverse, national sample of emergency department (ED) and hospital settings.

Primary Endpoints:

1. Emergency Department: The proportion of eligible children who receive systemic steroids within 60 minutes of ED arrival
2. Inpatient/Hospital: Mean length of hospital stay

Study Design:

This project will be implemented through an established quality improvement collaborative of hospitals across the United States, the Value in Inpatient Pediatrics Network (part of the American Academy of Pediatrics). A cluster randomized design will be employed. Group 1 hospitals will receive a multifaceted implementation strategy that includes: 1) a pathway implementation toolkit, 2) local multidisciplinary champions in the ED and inpatient settings, 3) audit and feedback, 4) educational seminars, and 5) practice facilitation (via teleconference). Group 2 will receive the same intervention with the addition of a mobile app pathway tool.

ELIGIBILITY:
Participant/Local champion Eligibility Criteria:

Inclusion Criteria:

* Working as a physician at the study site

Exclusion Criteria:

* None

Patient/child eligibility criteria:

Inclusion Criteria:

* Age 2-17 years
* Primary diagnosis of asthma

Exclusion Criteria:

* Transferred in from another inpatient facility
* Presence of a chronic medical condition that precludes pathway use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Hospital/Inpatient: Mean length of hospital stay | 1 year
Emergency Department: Proportion of eligible children who receive systemic steroids within 60 minutes of ED arrival | 1 year

SECONDARY OUTCOMES:
Hospital/Inpatient: Proportion of children with administration of bronchodilator via metered-dose inhaler early in hospitalization | 1 year
Hospital/Inpatient: Proportion of children screened for secondhand tobacco smoke exposure | 1 year
Hospital/Inpatient: Proportion of children who screen positive for secondhand tobacco smoke exposure whose caregivers are referred to smoking cessation resources | 1 year
Hospital/Inpatient: Proportion of children prescribed antibiotics at hospital discharge | 1 year
Hospital/Inpatient: Proportion of children with emergency department visits or readmissions to the hospital within 7 days | 1 year
Hospital/Inpatient: Proportion of children transferred to a higher level of care | 1 year
Emergency Department: Proportion of children who get an asthma exacerbation severity assessment at ED triage | 1 year
Emergency Department: Proportion of children who have chest radiographs performed | 1 year
Emergency Department: Proportion of children admitted to the hospital | 1 year
Emergency Department: Proportion of children transferred to a higher level of care | 1 year
Emergency Department: Mean length of emergency department stay | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sunitha V Kaiser, MD MSc, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No